CLINICAL TRIAL: NCT06597370
Title: Immunogenicity Induced by COVID-19 Vaccines in Mexican Population: mRNA Expression for IgG Anti-spike
Brief Title: Immunogenicity Induced by COVID-19 Vaccines in Mexican Population
Acronym: Vaccines COVID
Status: Completed | Type: Observational
Sponsor: National Polytechnic Institute, Mexico (Other)
Responsible Party: Principal Investigator, Modesto Gómez López, Immunogenicity induced by COVID-19 vaccines in Mexican population: mRNA expression for IgG anti-spike., National Polytechnic Institute, Mexico
Other Study IDs: CEI-01-2021
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: COVID-19 Vaccine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1: 20 persons who have received the Oxford/AstraZeneca vaccine (ChAdOx1 nCoV-19).
  Interventions: Other: Gene expression mRNA of IgG anti-spike
- Group 2: 20 persons who have received the vaccine Gamaleya National Center(Sputnik V)
  Interventions: Other: Gene expression mRNA of IgG anti-spike
- Group 3: 20 persons who have received the Pfizer/BioNTech vaccine (BNT162b2).
  Interventions: Other: Gene expression mRNA of IgG anti-spike
- Group 4: 20 persons who have received the Sinovac (CoronaVac) vaccine.
  Interventions: Other: Gene expression mRNA of IgG anti-spike

INTERVENTIONS:
Other: Gene expression mRNA of IgG anti-spike — b) Peripheral venous blood samples (3 ml per occasion) will be taken from all participants. They will be carried out on days 30,60 and 120 after completion of the COVID-19 vaccination schedule.
  c) Sample processing:
  * tRNA extraction from all samples.
  * cDNA synthesis
  * Real time PCR performance.

SUMMARY:
To determine the gene expression of anti-spike IgG through PCR-RT in patients vaccinated with the 4 types of vaccines available in Mexico Oxford/AstraZeneca (ChAdOx1 nCoV-19), Centro Nacional Gamaleya (Sputnik V), Pfizer/BioNTech (BNT162b2) and Sinovac (CoronaVac).

DETAILED DESCRIPTION:
80 subjects with full vaccination schedule will be included, 20 per group To know the gene expression of IgG anti-spike through PCR-RT in patients vaccinated with the 4 types of vaccines available in Mexico Oxford/AstraZeneca (ChAdOx1 nCoV-19), Centro Nacional Gamaleya (Sputnik V), Pfizer/BioNTech (BNT162b2) and Sinovac (CoronaVac).

ELIGIBILITY:
Inclusion Criteria:

1. - Mexican people.
2. - Over 18 years of age.
3. - With complete vaccination schedule against COVID-19.
4. - Allowing peripheral blood samples to be taken.
5. - To sign an informed consent form.
6. - To agree to participate in the protocol.

Exclusion Criteria:

1. - Persons with incomplete vaccination schedule against COVID-19.
2. - Persons who have 30 +/- 5 days of having completed the vaccination scheme against COVID-19.
3. - People under treatment with any immunosuppressive drug.
4. People who refuse to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mexican men and women over 18 years of age, vaccinated in the last 4 months
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Immunogenicity induced by COVID-19 vaccines in Mexican population | 4 months
  To characterize the immunogenicity induced by COVID-19 vaccines in Mexican population: mRNA expression for IgG anti-spike.

CONTACTS AND LOCATIONS:
Locations (1):
- Escuela Superior de Medicina, Instituto Politécnico Nacional, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Meyerowitz EA, Richterman A, Gandhi RT, Sax PE. Transmission of SARS-CoV-2: A Review of Viral, Host, and Environmental Factors. Ann Intern Med. 2021 Jan;174(1):69-79. doi: 10.7326/M20-5008. Epub 2020 Sep 17. PMID 32941052
- [Result] Pal M, Berhanu G, Desalegn C, Kandi V. Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2): An Update. Cureus. 2020 Mar 26;12(3):e7423. doi: 10.7759/cureus.7423. PMID 32337143
- [Result] Arya R, Kumari S, Pandey B, Mistry H, Bihani SC, Das A, Prashar V, Gupta GD, Panicker L, Kumar M. Structural insights into SARS-CoV-2 proteins. J Mol Biol. 2021 Jan 22;433(2):166725. doi: 10.1016/j.jmb.2020.11.024. Epub 2020 Nov 24. PMID 33245961
- [Result] Bourgonje AR, Abdulle AE, Timens W, Hillebrands JL, Navis GJ, Gordijn SJ, Bolling MC, Dijkstra G, Voors AA, Osterhaus AD, van der Voort PH, Mulder DJ, van Goor H. Angiotensin-converting enzyme 2 (ACE2), SARS-CoV-2 and the pathophysiology of coronavirus disease 2019 (COVID-19). J Pathol. 2020 Jul;251(3):228-248. doi: 10.1002/path.5471. Epub 2020 Jun 10. PMID 32418199
- [Result] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Result] Masters PS, Perlman S. Coronaviridae. 6th ed. Campos virología de, editor. Fields Virology. 2013. 825-58 p.
- [Result] Gonzalez JM, Gomez-Puertas P, Cavanagh D, Gorbalenya AE, Enjuanes L. A comparative sequence analysis to revise the current taxonomy of the family Coronaviridae. Arch Virol. 2003 Nov;148(11):2207-35. doi: 10.1007/s00705-003-0162-1. PMID 14579179
- [Result] Weiss SR, Navas-Martin S. Coronavirus pathogenesis and the emerging pathogen severe acute respiratory syndrome coronavirus. Microbiol Mol Biol Rev. 2005 Dec;69(4):635-64. doi: 10.1128/MMBR.69.4.635-664.2005. PMID 16339739
- [Result] Swelum AA, Shafi ME, Albaqami NM, El-Saadony MT, Elsify A, Abdo M, Taha AE, Abdel-Moneim AE, Al-Gabri NA, Almaiman AA, Saleh Al-Wajeeh A, Tufarelli V, Staffa VN, Abd El-Hack ME. COVID-19 in Human, Animal, and Environment: A Review. Front Vet Sci. 2020 Sep 4;7:578. doi: 10.3389/fvets.2020.00578. eCollection 2020. PMID 33102545
- [Result] Contini C, Di Nuzzo M, Barp N, Bonazza A, De Giorgio R, Tognon M, Rubino S. The novel zoonotic COVID-19 pandemic: An expected global health concern. J Infect Dev Ctries. 2020 Mar 31;14(3):254-264. doi: 10.3855/jidc.12671. PMID 32235085
- [Result] Majid S, Farooq R, Khan MS, Rashid S, Bhat SA, Wani HA, Qureshi W. Managing the COVID-19 Pandemic: Research Strategies Based on the Evolutionary and Molecular Characteristics of Coronaviruses. SN Compr Clin Med. 2020;2(10):1767-1776. doi: 10.1007/s42399-020-00457-z. Epub 2020 Aug 25. PMID 32864575
- [Result] Coronaviridae Study Group of the International Committee on Taxonomy of Viruses. The species Severe acute respiratory syndrome-related coronavirus: classifying 2019-nCoV and naming it SARS-CoV-2. Nat Microbiol. 2020 Apr;5(4):536-544. doi: 10.1038/s41564-020-0695-z. Epub 2020 Mar 2. PMID 32123347
- [Result] Lu H, Stratton CW, Tang YW. Outbreak of pneumonia of unknown etiology in Wuhan, China: The mystery and the miracle. J Med Virol. 2020 Apr;92(4):401-402. doi: 10.1002/jmv.25678. Epub 2020 Feb 12. No abstract available. PMID 31950516
- [Result] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. Addendum: A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Dec;588(7836):E6. doi: 10.1038/s41586-020-2951-z. No abstract available. PMID 33199918
- [Result] Park SE. Epidemiology, virology, and clinical features of severe acute respiratory syndrome -coronavirus-2 (SARS-CoV-2; Coronavirus Disease-19). Clin Exp Pediatr. 2020 Apr;63(4):119-124. doi: 10.3345/cep.2020.00493. Epub 2020 Apr 2. PMID 32252141

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT06597370/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT06597370/ICF_001.pdf